CLINICAL TRIAL: NCT03464175
Title: Influence of Respiratory Gases Conditioning on Aerosol Delivery During Invasive Ventilation: a Randomized Comparative Scintigraphic Study
Brief Title: Influence of Respiratory Gases Conditioning on Aerosol Delivery During Invasive Ventilation
Acronym: Aerovent-
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017/08NOV/508
Record Dates: First submitted 2018-03-04; First posted 2018-03-13 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Heated-humidifier left on during nebulization (Active Comparator)
  Interventions: Device: Aerogen Solo®; Device: Heated-humidified circuit
- Heated-humidifier turned off 30 minutes before nebulization (Active Comparator)
  Interventions: Device: Aerogen Solo®; Device: Heated-humidified circuit
- Use of a heat and moisture exchanger (HME) filter (Active Comparator)
  Interventions: Device: Aerogen Solo®; Device: Conventional dry ventilator circuit with HME filter
- Use of a dry ventilator circuit specific for aerosol therapy (Active Comparator)
  Interventions: Device: Aerogen Solo®; Device: Dry ventilator circuit specific for aerosol therapy

INTERVENTIONS:
Device: Aerogen Solo® — Aerosol particles are generated by a vibrating-mesh nebulizer specifically designed for mechanical ventilation
Device: Heated-humidified circuit — It will be left on during the transfer and the nebulization in group 1
  Arms: Heated-humidifier left on during nebulization
Device: Heated-humidified circuit — It will be turned off 30 minutes before the nebulization (nebulization ended max 45 minutes after turning off the heated-humidifier).
  Arms: Heated-humidifier turned off 30 minutes before nebulization
Device: Dry ventilator circuit specific for aerosol therapy — Streamlined components, specific position for the nebulizer at 30 cm of a V-shaped Y piece
  Arms: Use of a dry ventilator circuit specific for aerosol therapy
Device: Conventional dry ventilator circuit with HME filter — The nebulizer is placed between the filter and the endotracheal tube.
  Arms: Use of a heat and moisture exchanger (HME) filter

SUMMARY:
The intention is to enroll a specific sample of intubated patients. To compare the effect of respiratory gas conditioning on lung deposition and considering the well-known influences of lung pathology on lung deposition, intubated patients with healthy lungs will be included. Postoperative neurosurgery ventilated patients respond perfectly to this criteria. A previous study including 17 postoperative neurosurgery patients was performed in 2013 with a perfect collaboration between the ICU and the Department of Neurosurgery and Anesthesiology.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Postoperative neurosurgery intubated patients admitted for brain neurosurgery in the ICU (Intensive care neuro-traumatologic and Toxicologic)- With a healthy lung function.
* Signed and dated informed consent should be obtained in accordance of local regulations.

Exclusion Criteria:

* Spine neurosurgery
* History of cardiovascular and pulmonary disease
* Extubation immediately after surgery
* Modification of the allocated humidification technique before or during the nebulization (heated-humidifier deficiency or safety concern)
* Inaccurate quantification of aerosol deposition (i.e., artifacts or overlap of tracheal and pulmonary deposition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Quantity of aerosol deposition from the nebulizer reservoir to the subject. Measured by Planar scintigraphy. | 45 minutes
  % of the nominal dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universiataires Saint-Luc, Brussels, Belgium